CLINICAL TRIAL: NCT05878821
Title: Effect of Shockwave Therapy on Cervical Myofascial Pain Syndrome in Lactating Women
Brief Title: Effect of Shockwave Therapy on Cervical Myofascial Syndrome in Lactating Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Elham Shahat Hassan Baiuomy Ramadan, Lecturer of physical therapy Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/1004409
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cervical Myofascial Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Two groups,one group will be treated by shockwave therapy and postural correction exercise and other group will be treated by postural correction exercise
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postural correction exercise (Experimental): All women in both groups (A&B) will receive postural correction exercises which includes:
  A.mckenzie exercises:
  The exercise routine consists of seven types of movements,at static maximum strength, with 15_20 repetitions, holding each repetition for seven seconds.the subjects complete one 20-minutes set per day,three times a week for four weeks B.strengthening exercise targeted the periscapular muscles (Y to W,l to W), scapular retraction.strengthening exercises will be progressively performed for 3sets, with 10 to15 repetitions C.pectoralis flexibility on a foam roller.Hold for 5seconds and repeated 10 time s
  Interventions: Device: Shockwave
- Shockwave therapy (Experimental): All women in group (B) will receive shockwave therapy once a week for the duration of the trial (4 weeks)
  The dosage used will be as the following:
  Energy flux Density (EFD)=0,25 ml/mm2 Number of shocks=1000 shocks(kamel et al.,2020). Time:2-5minutes per session.
  Interventions: Device: Shockwave

INTERVENTIONS:
Device: Shockwave — Shockwave therapy session once a week for month 1000shock per session
  Other Names: Postural correction exercise

SUMMARY:
the aim of the study is to determine the effect of shockwave therapy on cervical myofascial pain syndrome in lactating women

DETAILED DESCRIPTION:
Neck and shoulder pain was 73,1%,one fourth of which occurred after birth.the most common area was the superior part of the trapezius.the symptoms of patients are pain, stiffness and limited range of motion (ROM).

ELIGIBILITY:
Inclusion Criteria:

* Multipara two months after labor.
* number of parity not more than 3.
* age range 25_35.BMI less than 35 Kg/m2

Exclusion Criteria:

* Diabetic women
* Women with malignancy
* Neck pain from other conditions such as(spinal
* instability, spinal fracture, spinal cord compression,inflammatory disease, spinal infection, congenital postural deformity

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 4 weeks
  Pain level will be assessed for both groups (A&B) before and after treatment program by using (VAS). scores are based on self-reported measures of symptoms that are recorded with a single hand written mark placed at one point along the length of a10 cm line."0 cm" means no pain."10cm" means maximum pain.
Pressure Algometer | 4 weeks
  Pain threshold for each woman in both groups (A&B) will be measured before and after the treatment program by using "Pressure Algometer" . The pressure pain threshold measurements for trapezius will be performed at mid-way between the seventh cervical vertebrae and acromial angle in limited area in the second and third quadrants (Barbero et al.' 2013).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No